CLINICAL TRIAL: NCT01408225
Title: Buckeye Surveillance, Contact, and Research for Multiple Myeloma and Amyloidosis
Brief Title: Ohio State University Multiple Myeloma and Amyloidosis Data Registry and Sample Resource
Acronym: B-SCR-MM
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Don Benson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-10115
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Plasma Cell Dyscrasias; Monoclonal Gammopathy of Undetermined Significance; AL Amyloidosis; Multiple Myeloma
Keywords: MGUS; Multiple Myeloma; Tissue Bank
MeSH Terms: conditions — Paraproteinemias; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis; Multiple Myeloma | interventions — Tissue Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — blood and bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: tissue banking — tissue procurement for this protocol will occur at the time of initial diagnosis, during routine follow-up, or at the time of relapse.

SUMMARY:
The investigators are researching patients with diseases of their plasma cells in order to improve their quality and length of life. The investigators have created a database of patient information, blood samples, and bone marrow tissue in order to achieve the following three goals:

* Surveillance: The investigators want to track what treatments patients get or don't get, how effective they are, how they feel, what complications they suffer, how long they stay in remission, and how long they live.
* Contact: Because myeloma and amyloidosis are rare, less than 700 patients are diagnosed in the state of Ohio each year, patients often feel they don't have accurate information. The investigators want to provide them access to our clinical team (both phone and email consultations, even office visits for patients that can come to Columbus) as well as information regarding informational events pertaining to your disease and local support groups.
* Research: Because nearly all myeloma and amyloid patients relapse and treatment is eventually unsuccessful, our focus is to develop more effective treatments that not only prolong life, but cure the disease. Periodically the investigators will inform them about clinical trials studying new drugs or treatment paradigms.

DETAILED DESCRIPTION:
The investigators propose to contact and interact with all patients with plasma cell dyscrasias in the State of Ohio (and all patients diagnosed or treated at Ohio State Medical Center) for both surveillance and research purposes in order to develop interventions targeted to decrease their morbidity and mortality.

ELIGIBILITY:
Inclusion:

Diagnosis of a plasma cell dyscrasia

Exclusion:

Prisoners are excluded from participation as they have no standard access to the Ohio State myeloma clinic and would impede the research objective of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated or diagnosed within the state of Ohio
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-03-17 (Actual); Primary Completion 2050-03 (Estimated); Study Completion 2050-03 (Estimated)

PRIMARY OUTCOMES:
Develop a data and sample resource that can be used to facilitate research with the ultimate goal of reducing the morbidity and/or mortality of patients diagnosed or living with Multiple Myeloma in the state of Ohio | up to 3 years

SECONDARY OUTCOMES:
Surveillance | up to 3 years
  Establish a database of myeloma patients diagnosed or living in the state of Ohio to track myeloma disease course, patient reported outcomes, morbidity, and patient survival.
Contact | up to 3 years
  Provide two-way communication with patients by providing information regarding multiple myeloma, local support groups, and standard of care procedures through active contact procedures
Research | up to 3 years
  Offer patients, and occasionally spouses and family members, the opportunity to participate in tissue banking, observational, patient reported outcomes, and therapeutic clinical trials for their plasma cell dyscrasia.

CONTACTS AND LOCATIONS:
Overall Officials: Don Benson, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Khalife J, Ghose J, Martella M, Viola D, Rocci A, Troadec E, Terrazas C, Satoskar AR, Gunes EG, Dona A, Sanchez JF, Bergsagel PL, Chesi M, Pozhitkov A, Rosen S, Marcucci G, Keats JJ, Hofmeister CC, Krishnan A, Caserta E, Pichiorri F. MiR-16 regulates crosstalk in NF-kappaB tolerogenic inflammatory signaling between myeloma cells and bone marrow macrophages. JCI Insight. 2019 Nov 1;4(21):e129348. doi: 10.1172/jci.insight.129348. PMID 31593552